CLINICAL TRIAL: NCT01966783
Title: Randomized, Double-blind, Multicentre Study to Compare the Efficacy and Safety of Budesonide Versus Mesalazine Suppository Versus a Combination Therapy of Budesonide/Mesalazine Suppositories in Patients With Acute Ulcerative Proctitis
Brief Title: Budesonide vs. Mesalazine vs. Budesonide/Mesalazine Suppository Combination Therapy in Acute Ulcerative Proctitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUS-2/UCA; 2012-003362-41 (EudraCT Number)
Record Dates: First submitted 2013-10-09; First posted 2013-10-22 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Proctitis
MeSH Terms: conditions — Proctitis | interventions — Budesonide; Suppositories; Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Budesonide dosage 1 (Experimental): Budesonide 2 mg suppository
  Interventions: Drug: Budesonide 2 mg suppository
- Budesonide dosage 2 (Experimental): Budesonide 4 mg suppository
  Interventions: Drug: Budesonide 4 mg suppository
- Mesalazine (Active Comparator): Mesalazine 1g suppository
  Interventions: Drug: Mesalazine 1 g suppository
- Combination (Experimental): Budesonide 2 mg suppository/Mesalazine 1 g suppository
  Interventions: Drug: Budesonide 2 mg suppository/Mesalazine 1 g suppository

INTERVENTIONS:
Drug: Budesonide 2 mg suppository — per day
  Arms: Budesonide dosage 1
Drug: Budesonide 4 mg suppository — per day
  Arms: Budesonide dosage 2
Drug: Mesalazine 1 g suppository — per day
  Arms: Mesalazine
Drug: Budesonide 2 mg suppository/Mesalazine 1 g suppository — per day
  Arms: Combination

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of budesonide suppository for the treatment of acute ulcerative proctitis.

ELIGIBILITY:
Inclusion Criteria:

* Active ulcerative proctitis
* Diagnosis confirmed by endoscopy
* Established disease or new diagnosis

Exclusion Criteria:

* Crohn's disease, indeterminate colitis, ischemic colitis, radiation colitis, diverticular assoc. colitis, microscopic colitis
* Presence of proctitis of a different origin
* Prior bowel resection
* Presence of symptomatic organic disease of the gastrointestinal tract
* Asthma, tuberculosis, cardiovascular disease, diabetes mellitus, osteoporosis, active peptic ulcer disease, glaucoma, cataract, infection if careful medical monitoring is not ensured
* Local intestinal infection
* Abnormal hepatic or renal function
* Oral/rectal/intravenous corticosteroids therapy
* Existing or intended pregnancy or breast-feeding
* Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Resolution of clinical symptoms | 8 weeks
  Symptoms as reported in the diary

SECONDARY OUTCOMES:
Rate of clinical and endoscopic remission | 8 weeks
  Symptoms as reported in the diary, ulcerative colitis-disease activity index
Rate of improvement | 8 weeks
  Symptoms as reported in the diary, ulcerative colitis-disease activity index
Rate of patients with clinical remission | 8 weeks
  Symptoms as reported in the diary, ulcerative colitis-disease activity index
Rate of patients with endoscopic remission | 8 weeks
  Ulcerative colitis-disease activity index

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kruis, Professor, Principal Investigator — Evang. Krankenhaus Kalk, Medical Department; Britta Siegmund, Professor, Principal Investigator — Charité-Campus Benjamin Franklin Universitätsmedizin Berlin
Locations (2):
- Germany (2):
  - Charité-Campus Benjamin Franklin Universitätsmedizin Berlin, Berlin
  - Evang. Krankenhaus Kalk, Medical Department, Cologne

REFERENCES:
- [Result] Kruis W, Neshta V, Pesegova M, Alekseeva O, Andreev P, Datsenko O, Levchenko O, Abdulkhakov S, Lozynskyy Y, Mostovoy Y, Soloviev K, Dorofeyev AE, Vieth M, Stiess M, Greinwald R, Mohrbacher R, Siegmund B. Budesonide Suppositories Are Effective and Safe for Treating Acute Ulcerative Proctitis. Clin Gastroenterol Hepatol. 2019 Jan;17(1):98-106.e4. doi: 10.1016/j.cgh.2018.04.027. Epub 2018 Apr 24. PMID 29702300